CLINICAL TRIAL: NCT00658164
Title: Effect of Iron Depletion by Phlebotomy Plus Lifestyle Changes vs. Lifestyle Changes Alone on Liver Damage in Patients With Nonalcoholic Fatty Liver Disease With Increased Iron Stores
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Fondazione Ospedale Maggiore Policlinico Mangiagalli e Regina Elena, Prof. Silvia Fargion
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111.2007
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2007-07

CONDITIONS: Nonalcoholic Fatty Liver Disease
Keywords: Nonalcoholic fatty liver disease associated with increased iron stores
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Iron depletion treatment

INTERVENTIONS:
Other: Iron depletion treatment — Effect of iron depletion by phlebotomy plus lifestyle changes vs. lifestyle changes alone on liver damage in patients with nonalcoholic fatty liver disease with increased iron stores

SUMMARY:
Patients will be randomized to lifestyle changes alone or lifestyle changes associated with iron depletion.

Iron depletion will be achieved by removing 350 cc of blood every 10-15 days according to baseline hemoglobin values and venesection tolerance, until ferritin < 30 ng/ml and transferrin saturation < 25%. Weekly phlebotomies will be allowed for carriers of the C282Y HFE mutation. Smaller phlebotomies (250 cc) will be allowed for carriers of beta-thalassaemia trait. Maintenance phlebotomies (as much as required) will then be instituted to keep iron stores depleted (ferritin < 50 ng/ml and transferrin saturation < 25%, MCV <85 fl). Before starting treatment, patients will undergo ECG, and in the presence of hyperglycemia or hypertension also echocardiography (see exclusion criteria).

Change in diabetes medication dosage or start of new therapy will be allowed for HbA1C values <6% or ≥ 7%. According to accepted criteria, previously untreated patients should be treated with metformin. If possible, newly diagnosed hypertension should be treated with Ace-inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 < 75 years
* Ferritin > 250 ng/ml and/or stainable iron at biopsy
* NAS ≥ 2 and/or NAS 1 and stage≥1 at liver histology
* Willingness to maintain diet and exercise during the full course of the study
* Written informed consent to participate to the study and to have the specific genetic tests performed
* Ability to comply with all study requirements

Exclusion Criteria:

* Pregnant or lactating female
* Diagnosis of or a history of:
* Type 1 diabetes, diabetes that is a result of pancreatic injury, or secondary forms of diabetes, e.g. Cushing's syndrome or acromegaly
* Acute metabolic complication such as ketoacidosis or hyperosmolar state within the past 6 months
* Alcohol consumption > 20 g/day for females and > 30 g/day for males
* BMI ≥ 35 Kg/ m2
* Other liver disease such as viral hepatitis, autoimmune hepatitis, Wilson disease, as defined by ceruloplasmin below normal limits and liver histology consistent with Wilson disease. Alpha-1-antitrypsin deficiency as defined by alpha-1-antitrypsin level less than 80 mg/dl or PiZ/PiZ or PiZ/PiS genotype. *Hemochromatosis, as defined by homozygosity for the C282Y HFE mutation or compound heterozygosity for C282Y/H63D mutations or Hepatic Iron Index ≥ 1.9.
* Advanced liver disease (Child B/C cirrhosis), portal hypertension, hepatocellular carcinoma.
* Congestive heart failure (NYHA I-IV) and unstable ischemic heart disease, systolic dysfunction (ejection fraction < 45%)
* Any of the following ECG abnormalities: II or III degree Atrial Ventricular *Block, QT>500msec, repolarization defect suggestive of ischemia
* Malignancy within the last 5 years
* Serum creatinine levels > 1.5 mg/dl males, > 1.4 mg/dl females
* TSH outside of normal range
* Use of drugs known to induce NAFLD: corticosteroids, methotrexate, zidovudine, amiodarone, GH, estrogens, tamoxifene, tetracycline
* Lipodystrophy, dysbetalipoproteinemia, inflammatory bowel disease, HIV infection
* Basal hemoglobin levels < 11 g/dl

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
To determine in a 24 month controlled study whether iron depletion by phlebotomy improves insulin sensitivity, and thereby reduces hepatic steatosis and inflammation in subjects with nonalcoholic steatohepatitis | 24 months

SECONDARY OUTCOMES:
To assess the effect of iron depletion on glucose tolerance status. Glucose tolerance will be determined by OGTT in subjects without type 2 diabetes (T2D), and by HbA1c levels and the change in dosage of pharmacological therapy in those with T2D. | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- U.O. Medicina Interna 1/B, Milan, Italy